CLINICAL TRIAL: NCT04016818
Title: Pilot Study of a Breast-Dedicated PET Camera With 1 Millimeter Spatial Resolution
Brief Title: Pilot Breast-Dedicated PET Camera With 1 Millimeter Spatial Resolution
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-50877; BRS0102 (Other: OnCore); IRB-50877 (Other: Stanford IRB)
Record Dates: First submitted 2019-07-02; First posted 2019-07-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- 18-F FDG Study using Breast-Dedicated PET Camera (Experimental): Breast-Dedicated PET Camera will be used with standard PET 18-F FDG tracer dose
  Interventions: Drug: 18F-FDG; Device: Breast-dedicated PET camera

INTERVENTIONS:
Drug: 18F-FDG — Participant will be injected IV (intravenously) with 10 ± 2 mCi of 18F-FDG.
  Other Names: 18F-fluorodeoxiglucose; 18F-FDG radiotracer
Device: Breast-dedicated PET camera — Breast-dedicated PET camera designed by Stanford satellite radiochemistry facility

SUMMARY:
This is a research study of a novel, "breast-dedicated" positron emission tomography (PET) camera with 1 millimeter spatial resolution. The main goal of the study is for the personnel to understand practical and logistical issues with using the camera in the clinic

DETAILED DESCRIPTION:
Primary Objective To obtain initial experience using the novel, breast-dedicated PET camera design in the breast imaging clinic.

Secondary Objectives To understand, given the 10-fold higher sensitivity of this novel camera, how low we can go with administered tracer dose, and, given the >100-fold better volumetric spatial resolution, understand the achievable image quality.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed breast cancer measuring ≥ 5 mm on mammogram or ultrasound.
* Prior diagnostic imaging test(s) with another modality such as MRI, CT, or x-ray mammography (or other applicable imaging modalities) within 60 days prior to the study date.
* Documented written informed consent document.

Exclusion Criteria:

* 1. Additional condition, or extenuating circumstance that, in the opinion of the investigator, may interfere with study compliance.
* Known allergies to FDG
* Pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Image quality with the breast-dedicated PET camera | 1 day
  Feasibility of the pilot breast-dedicated PET camera will be assessed on the basis of whether acceptable images are obtained. Images will be assessed and graded as 1 of 3 quality ratings: excellent, good, and poor. The outcome will be reported as the number of images that are excellent, good, and poor, a number without dispersion.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy B DeMartini, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No